CLINICAL TRIAL: NCT04542135
Title: Double-blind, Randomized Phase II Clinical Trial of Sulindac for Reducing Breast Density in Postmenopausal Women at Risk of Developing Breast Cancer
Brief Title: Sulindac and Breast Density in Women at Risk of Developing Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alison Stopeck (Other)
Collaborators: Medical University of South Carolina (Other); Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor-Investigator, Alison Stopeck, Principal Investigator, Stony Brook University
Organization: Stony Brook University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STOP-BC Trial
Record Dates: First submitted 2020-08-27; First posted 2020-09-09 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: Breast Density
MeSH Terms: conditions — Breast Neoplasms | interventions — Sulindac

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sulindac (Active Comparator): sulindac 150 mg
  Interventions: Drug: Sulindac Pill
- Placebo (Placebo Comparator): placebo pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sulindac Pill — Randomized participants will receive either 150 mg oral sulindac twice daily.
  Arms: Sulindac
Drug: Placebo — placebo pills twice daily
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine if sulindac at a dose of 150 mg twice a day for 12 months reduces breast density in postmenopausal women at elevated risk of breast cancer when compared to a placebo control.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤70 years
2. Subject must be postmenopausal.
3. Must have at least one healthy normal appearing breast (no prior diagnosis of invasive cancer, radiation or prosthetics). Prior biopsies are acceptable.
4. Must have dense breasts
5. Must be at elevated risk for developing breast cancer by abnormal pathological findings, family history, or genetic predisposition
6. A negative fecal occult blood test
7. Normal organ function
8. Hormonal therapy with aromatase inhibitors is allowed

Exclusion Criteria:

1. Daily aspirin or other daily anti inflammatory use.
2. Known intolerance to anti inflammatory.
3. Use of any selective estrogen receptor modulator therapy (e.g., tamoxifen, raloxifene) within past 12 months
4. Gastrointestinal, bleeding or coagulation, cardiovascular disorders.
5. Diabetes requiring insulin therapy.
6. Current regular smoker.
7. History of claustrophobia or inability to undergo imaging in a closed magnetic resonance imaging.
8. Cardiac pacemaker, cochlear implants, magnetic surgical clips or prostheses that would preclude MRI.
9. Uncontrolled hypertension.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
Change in percent breast density by MRI between treatment arms | 12 months

SECONDARY OUTCOMES:
Change in percent breast density by MRI between treatment arms | 6 months
Changes in in percent breast density by MRI within and between treatment arms, stratified by use of aromatase inhibitors | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alison S Stopeck, MD, Principal Investigator — Stony Brook University; Patricia A Thompson-Carino, PhD, Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - Cedars Sinai - Cancer, Los Angeles, California
  - Stony Brook University Cancer Center, Stony Brook, New York

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data to non study related researchers.